CLINICAL TRIAL: NCT00749177
Title: Blending Two Worlds: Traditional Aboriginal Healing Strategies for Depression and Anxiety. Possible Options for Children, Youth and Families
Brief Title: Blending Two Worlds: Traditional Aboriginal Healing Strategies for Depression and Anxiety
Acronym: B2W
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator left program: unable to recruit a replacement
Sponsor: Fraser Health (Other)
Collaborators: Ministry of Children and Family Development, British Columbia (Other)
Responsible Party: Principal Investigator, Debbie Thompson, Clinical Pharmacy Specialist, Fraser Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FHA-MHA-B2W
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Anxiety; Depression
Keywords: traditional healing; anxiety; depression; aboriginal; children; youth
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): Traditional Healing arm Provides Traditional Healing options only
  Interventions: Other: Traditional Healing options
- 3 (Active Comparator): Traditional Healing and usual standard of care arm Subjects will access both treatment options
  Interventions: Other: Traditional Healing options
- 1 (Active Comparator): Treatment as usual
  Interventions: Other: Traditional Healing options

INTERVENTIONS:
Other: Traditional Healing options — Dream work, energy healing, healing circles, pipe ceremonies, self care, smudging, sweat lodges and traditional learning.

SUMMARY:
1. Purpose

   1. Provide a culturally sensitive and supportive treatment environment for children, youth and families in the aboriginal community experiencing stress, anxiety and depression.
   2. Gain insight into understanding of the role of Traditional Healing options provided by Aboriginal Healers and Helpers in the management of stress, anxiety and depression.
   3. Encourage Aboriginal and First Nation clients to seek treatment earlier from a culturally supportive system.
2. Hypothesis

This will be a descriptive hypothesis generating research project, however it is anticipated that members of the Aboriginal community experiencing stress, anxiety and depression may experience improved care and outcomes if their treatment includes traditional healing methods. A number of measures of subject and treatment characteristics, stress, anxiety and depression will provide the foundation for triangulation of outcomes in order to describe the impact of the various treatment options (standard care, Traditional Healing, combined standard care and Traditional Healing).

DETAILED DESCRIPTION:
Aboriginal clients, including first nation youth, may not be confident or comfortable with the standard treatments offered by the current Mental Health environment. Incorporating traditional aboriginal healing methods such as dream work, energy healing, healing circles, pipe ceremonies, self care, smudging, sweat lodge and traditional learning into standard practice will provide a culturally sensitive and supportive environment for children, youth and families experiencing stress, anxiety and depression.

It is believed that Aboriginal and First Nation clients that access treatment options consistent with cultural beliefs will be encouraged to seek treatment earlier and will experience improved care and outcomes.

In addition, the improved understanding of the role of traditional healing methods provided by Aboriginal Healers and Helpers in the management of these disorders will help clinicians incorporate these practices in the management of anxiety and depression

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents (less than 18 years of age)and families with anxiety and/or depression attending the Surrey North Child and Youth Mental Health Team.

Exclusion Criteria:

* Subjects with severe anxiety or depression requiring intervention (i.e. hospitalization) or have a past or present history of suicide attempt. Subjects with special needs including medical contraindications (i.e. medical conditions including pregnancy), brain injury, developmental disability or fetal alcohol syndrome). Those subjects unwilling or unable to participate in a Traditional Healing options.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Provide Aboriginal and First Nation youth and their families with treatment options consistent with cultural beliefs. Improving outcomes in the management of anxiety and depression. | Within one year

SECONDARY OUTCOMES:
1. Encourage Aboriginal and First Nation clients to seek treatment earlier from a culturally supportive system. 2. Validate the benefit of traditional diet and healing methods in the treatment of stress, anxiety and depression | Within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Thompson, BScPharm, BCPP, PharmD, Principal Investigator — Fraser Health
Locations (1):
- Child and Youth Mental Health, Surrey North, Surrey, British Columbia, Canada

REFERENCES:
- [Background] Hunter L, Logan J, Barton S, Goulet JG. Linking aboriginal healing traditions to holistic nursing practice. J Holist Nurs. 2004 Sep;22(3):267-85. doi: 10.1177/0898010104266750. PMID 15296579
- [Background] Dapice AN. The medicine wheel. J Transcult Nurs. 2006 Jul;17(3):251-60. doi: 10.1177/1043659606288383. PMID 16757664
- [Background] Struthers R, Hodge FS. Sacred tobacco use in Ojibwe communities. J Holist Nurs. 2004 Sep;22(3):209-25. doi: 10.1177/0898010104266735. PMID 15296576
- [Background] Buehler JA. Traditional Crow Indian health beliefs and practices. Toward a grounded theory. J Holist Nurs. 1992 Mar;10(1):18-33. doi: 10.1177/089801019201000104. PMID 1293200
- [Background] Zubek EM. Traditional Native healing. Alternative or adjunct to modern medicine? Can Fam Physician. 1994 Nov;40:1923-31. PMID 7841824
- [Background] Buchwald D, Beals J, Manson SM. Use of traditional health practices among Native Americans in a primary care setting. Med Care. 2000 Dec;38(12):1191-9. doi: 10.1097/00005650-200012000-00006. PMID 11186298